CLINICAL TRIAL: NCT03165981
Title: A Prospective, Randomized, Open-label Clinical Trial to Assess Fever Following Simultaneous Versus Sequential Administration of PCV13, DTaP Vaccine and IIV in Young Children
Brief Title: Fever After Simultaneous Versus Sequential Vaccination in Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00082484; 200 2012 53663 0009 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Results first posted 2019-02-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Fever After Vaccination; Fever; Febrile Seizure
Keywords: Influenza vaccine; fever following vaccination; PCV13 vaccine; DTaP vaccine; pneumococcal vaccine
MeSH Terms: conditions — Fever; Seizures, Febrile; Influenza, Human | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Simultaneous vaccination arm (Other): In the study arm, subjects will receive PCV13, DTaP and IIV vaccines during visit 1. Approximately 2 weeks later, subjects will receive a health education visit without vaccination during study visit 2.
  Interventions: Biological: PCV13; Biological: DTaP; Biological: IIV
- Sequential vaccination arm (Other): In the study arm, subjects will receive PCV13 and DTaP during study visit 1. Approximately 2 weeks later, subjects will receive the IIV vaccine during study visit 2.
  Interventions: Biological: PCV13; Biological: DTaP; Biological: IIV

INTERVENTIONS:
Biological: PCV13 — ACIP Recommended vaccine
  Other Names: 13-valent Conjugate Pneumococcal Vaccine
Biological: DTaP — ACIP Recommended vaccine
  Other Names: Diphtheria, Tetanus, and Acellular Pertussis Vaccine
Biological: IIV — ACIP Recommended vaccine
  Other Names: Quadrivalent Inactivated Influenza Vaccine; IIV4; Flu Vaccine

SUMMARY:
A prospective, randomized open-label clinical trial that will be conducted during the 2017-2018 influenza season. During the 2017-2018 season, approximately 280 children will be enrolled at Duke University Medical Center and Kaiser Permanente Northern California. Eligible children will be randomized to receive simultaneous or sequentially administered US licensed PCV13, US-licensed DTaP vaccine, and US-licensed inactivated influenza vaccine (IIV). Children in the simultaneous group will receive PCV13, DTaP, and IIV vaccines at Visit 1, and then return for a health education visit without vaccination about 2 weeks later (Visit 2). Children in the sequential group will receive both PCV13 and DTaP without IIV at Visit 1, and then will receive IIV and health education about 2 weeks later (Visit 2). Parents will record the occurrence of fever, solicited adverse events, medical care utilization, and receipt of antipyretics over 8 days following Visit 1 and Visit 2. In addition, febrile seizures and serious adverse events will be recorded for the entire study period (from enrollment through 8 days following the Visit 2) as determined through parental report and chart review. Parental perceptions about their child's vaccine schedule will be assessed on the 8th day following Visit 2.

ELIGIBILITY:
Inclusion Criteria:

1. 12 through 16 months of age (i.e. from the 1-year birthday until the day before 17 months of age) at the time of vaccination
2. Stable health as determined by investigator's clinical examination and assessment of child's medical history
3. Has received all immunizations recommended by Advisory Committee for Immunization Practices (ACIP) during the first year of life with the exception of rotavirus and influenza vaccines.
4. The parent(s)/ legally authorized representative(s) LAR(s) intend for the child to receive DTaP and PCV13 in addition to this season's IIV
5. The parent(s)/LAR(s) must be willing and capable of providing permission for their child to participate through the written informed consent process
6. The parent(s)/LAR(s) must be able to comply with the requirements of the protocol (e.g., completion of the memory aid (either electronic or paper diary), return for follow-up visits, respects intervals between the visits and have telephone access.
7. The parent(s)/LAR(s) must be English speaking
8. The parent(s)/LAR(s) must agree to sign a medical release for the child so that study personnel may obtain medical information about the child's health (if needed)

Exclusion Criteria:

1. History of any seizure (including febrile seizure) in the child or a febrile seizure in a first degree relative
2. Has already completed influenza vaccination during the current season per ACIP recommendations
3. Receipt of more than 3 previous doses of DTaP
4. Received the 3rd dose of DTaP within 6 months of Visit 1
5. Receipt of more than 3 previous doses of PCV13
6. Received the 3rd dose of PCV13 within 8 weeks of Visit 1
7. History of a severe allergic reaction (e.g. anaphylaxis) to a previous dose of any influenza, diphtheria toxoid-, tetanus toxoid-, or pertussis-containing vaccine, or pneumococcal vaccine.
8. History of a severe allergic reaction (e.g., anaphylaxis) to any component (including egg protein) of any of the three vaccines used in this study; or a latex allergy.
9. History of Guillain-Barré syndrome within 6 weeks following a prior dose of influenza, DTaP, or tetanus toxoid containing vaccine
10. History of a progressive neurologic disorder
11. History of encephalopathy within 7 days of a previous pertussis-containing vaccine
12. History of collapse within 3 days after a prior dose of DTaP
13. Received any other licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to Visit 1
14. Received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 28 days prior to Visit 1, or expects to receive an experimental/investigational agent during the study period (up to 8 days after visit 2)
15. A moderate to severe acute illness within 72 hours of Visit 1
16. A reported temperature greater than or equal to 100.4°F (38.0°C) within 72 hours prior enrollment or a temperature (measured by temporal artery thermometer) greater than or equal to 100.4°F (38.0°C) at the time of enrollment
17. Receipt of an antipyretic medication (acetaminophen or ibuprofen) within 24 hours prior to enrollment
18. Parent(s)/LAR is planning to administer a prophylactic antipyretic or medication on the day of, and/or within 7 days following Visit 1 or Visit 2
19. Long term (at least 14 consecutive days) oral corticosteroids (prednisone 2 mg/kg/day or equivalent other glucocorticoid), any parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immune-modifying drugs or immunosuppressants within the preceding 6 months prior to Visit 1
20. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and or their provider's routine physical examination
21. Has an active neoplastic disease, a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants.
22. Unable to receive an intramuscular injection in the thigh
23. Any condition deemed by the investigator to place the child at increased risk as a result of their participation in the study
24. Any child or grandchild of a study investigator or study team member

Ages: 12 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel B Walter, MD, MPH, Principal Investigator — Duke University; Karen Broder, MD, Principal Investigator — Centers for Disease Control and Prevention; Nicola Klein, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Kaiser Permanente Northern California, Oakland, California
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walter EB, Klein NP, Wodi AP, Rountree W, Todd CA, Wiesner A, Duffy J, Marquez PL, Broder KR. Fever After Influenza, Diphtheria-Tetanus-Acellular Pertussis, and Pneumococcal Vaccinations. Pediatrics. 2020 Mar;145(3):e20191909. doi: 10.1542/peds.2019-1909. Epub 2020 Feb 6. PMID 32029684

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Started (Intent-to-treat Population: enrolled, randomized and received at least one study vaccine at V1) | 110 | 111
Per Protocol Population (Excludes those w/o valid temperature data on D1-2 following V1-2 or with major protocol violations) | 99 | 107
Completed | 99 | 107
Not Completed | 11 | 4

BASELINE CHARACTERISTICS:
Population: Per Protocol Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm | Total
Number analyzed (Participants) | 99 | 107 | 206
Age, Continuous [Median (Full Range); unit: Months] | 14.1 [12.0 to 16.6] | 14.8 [12.0 to 16.9] | 14.7 [12.0 to 16.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 55 | 103
  Male | 51 | 52 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 22 | 43
  Not Hispanic or Latino | 78 | 85 | 163
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 9 | 16
  Asian | 6 | 11 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 10 | 6 | 16
  White | 52 | 57 | 109
  More than one race | 18 | 19 | 37
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 99 | 107 | 206
Insurance [Count of Participants; unit: Participants]
  Any Private | 63 | 84 | 147
  Public | 18 | 10 | 28
  None | 18 | 13 | 31
Number of Children Living in Home [Median (Full Range); unit: Children] | 2 [1 to 7] | 2 [1 to 5] | 2 [1 to 7]
Day Care [Count of Participants; unit: Participants]
  Full-time (4-5 days/weeks) | 22 | 34 | 56
  Part-time (3 or less/weeks) | 17 | 16 | 33
  None | 60 | 57 | 117
Gestational Age in Weeks [Median (Full Range); unit: Weeks] | 39 [34 to 42] | 39 [34 to 42] | 39 [34 to 42]
Birth Weight in Pounds [Median (Full Range); unit: Pounds] | 7.25 [4.69 to 10.31] | 7.13 [3.50 to 10.75] | 7.13 [3.50 to 10.75]
Receipt of 1st or Only Dose of Influenza Vaccine for the Season [Count of Participants; unit: Participants] | 90 | 102 | 192
Receipt of 2nd Dose of Influenza Vaccine for the Season [Count of Participants; unit: Participants] | 9 | 5 | 14
Receipt of Concomitant Vaccine [Count of Participants; unit: Participants] | 87 | 98 | 185

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fever Following Vaccination
Description: Proportion of children with fever (temperature ≥ 38.0°C or ≥ 100.4°F) on day 1 and/or day 2 following Visit 1 and/or Visit 2.
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 8 | 10
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = 0.7588, Mantel Haenszel; Mantel Haenzel is stratified by site; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.36 to 2.10] — RR is adjusted by site

2. Secondary Outcome: Number of Participants With Fever Visit 1
Description: Proportion of children with fever (temperature ≥ 38.0°C or ≥ 100.4°F) on day 1 and/or day 2 following Visit 1
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 8 | 9
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = .9412, Mantel Haenszel; Mantel Haenzel is stratified by site; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.39 to 2.40] — RR is adjusted by site

3. Secondary Outcome: Number of Participants With Fever Visit 2
Description: Proportion of children with fever (temperature ≥ 38.0°C or ≥ 100.4°F) on day 1 and/or day 2 following Visit 2
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 0 | 1
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = 0.3408, Mantel Haenszel; Mantel Haenzel is stratified by site

4. Secondary Outcome: Number of Participants With Grade 2 and/or 3 Fever Following Visit 1
Description: Proportions of children with moderate/severe fever (Grade 2 and/or 3) on day 1 and/or day 2 following Visit 1. (Moderate/severe fever: ≥ 38.6°C or ≥ 101.4°F)
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 4 | 5
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = 0.8325, Mantel Haenszel; Mantel Haenzel is stratified by site; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.24 to 3.13] — RR is adjusted by site

5. Secondary Outcome: Number of Participants With Grade 2 and/or 3 Fever Following Visit 2
Description: Proportions of children with moderate/severe fever (Grade 2 and/or 3) on day 1 and/or day 2 following Visit 2.
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 0 | 1
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = 0.3408, Mantel Haenszel; Mantel Haenzel is stratified by site

6. Secondary Outcome: Number of Participants With Grade 2 and/or 3 Following Visit 1 and Visit 2
Description: Proportions of children with moderate/severe fever (Grade 2 and/or 3) on day 1 and/or day 2 following Visit 1 and Visit 2 combined.
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 4 | 6
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = 0.6101, Mantel Haenszel; Mantel Haenzel is stratified by site; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.21 to 2.48] — RR is adjusted by site

7. Secondary Outcome: Duration of Fever - Visit 1
Description: Average number of consecutive days of fever (temperature ≥ 38.0°C or ≥ 100.4°F) per subject for fever starting on day 1 or 2 following Visit 1. Note: fever starting on day 1 or 2 could continue through day 8.
Time Frame: 8 days post administration
Population: Per Protocol Population
Measure: Mean (Full Range); unit: Fever Days
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Fever Days | 1.3 [1 to 2] | 1.4 [1 to 3]
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = 0.848, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Duration of Fever - Visit 2
Description: Average number of consecutive days of fever (temperature ≥ 38.0°C or ≥ 100.4°F) per subject for fever starting on day 1 or 2 following Visit 2. Note: fever starting on day 1 or 2 could continue through day 8.
Time Frame: 8 days post administration
Population: Per Protocol Population
Measure: Mean (Full Range); unit: Fever Days
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Fever Days | 0 [0 to 0] | 3 [3 to 3]

9. Secondary Outcome: Duration of Fever - Visit 1 and 2 Combined
Description: Average number of consecutive days of fever (temperature ≥ 38.0°C or ≥ 100.4°F) per subject for fever starting on day 1 or 2 following and Visit 1 and Visit 2 combined. Note: fever starting on day 1 or 2 could continue through day 8.
Time Frame: 8 days post administration
Population: Per Protocol Population
Measure: Mean (Full Range); unit: Fever Days
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Fever Days | 1.3 [1 to 2] | 1.6 [1 to 3]
Statistical Analysis 1: Comparison: Simultaneous Vaccination Arm vs Sequential Vaccination Arm; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of Participants With Medical Care Utilization - Visit 1
Description: Proportion of children with medical care utilization (telephone call, medical office visit, emergency department visit, or hospital admission) for fever on day 1 and/or day 2 following Visit 1.
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Medical Care Utilization - Visit 2
Description: Proportion of children with medical care utilization (telephone call, medical office visit, emergency department visit, or hospital admission) for fever on day 1 and/or day 2 following Visit 2.
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Medical Care Utilization - Visit 1 and 2 Combined
Description: Proportion of children with medical care utilization (telephone call, medical office visit, emergency department visit, or hospital admission) for fever on day 1 and/or day 2 following Visit 1 and Visit 2 combined.
Time Frame: 2 days post administration
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 99 | 107
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 8 days post Visit 2.
Description: All-cause mortality, serious adverse events, and other AEs exceeding a frequency threshold of 1% (febrile seizure only) were collected and reported. Per protocol, the only AE collected was febrile seizure.
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/99 | 1/107
Other Adverse Events (participants affected / at risk) | 0/99 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous Vaccination Arm (N=99) | Sequential Vaccination Arm (N=107)
Dehydration (General disorders) | 0 (0) | 1 (1) — Subject presented with fever, upper respiratory symptoms, decreased oral intake and dehydration 13 days after Visit 1. The SAE was considered unrelated to vaccination by the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03165981/Prot_SAP_000.pdf